CLINICAL TRIAL: NCT04538105
Title: Preoperative Fluoroscopy Guided Hip Articular Branch Blocks and Analgesic Outcomes Following Hip Arthroscopy: A Randomized, Controlled Trial
Brief Title: Preoperative Fluoroscopy Guided Hip Articular Branch Blocks and Analgesic Outcomes Following Hip Arthroscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study cancelled
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Tolga Suvar, MD, Principle Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20051404
Record Dates: First submitted 2020-08-17; First posted 2020-09-03 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Surgery, Arthroscopic; Analgesia; Pain, Acute
Keywords: hip arthroscopy; articular branch block
MeSH Terms: conditions — Agnosia; Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Injection (Sham Comparator): 20cc of Normal Saline 0.9%
  Interventions: Other: Control
- Articular Branch Block (ABB) (Experimental): 20cc of 0.5% Bupivacaine with epinephrine 1:200,000
  Interventions: Other: Articular Branch Block (ABB)

INTERVENTIONS:
Other: Control — Saline Articular Nerve Branch Block
  Arms: Sham Injection
Other: Articular Branch Block (ABB) — 0.5% Bupivacaine with epinephrine 1:200,000 (Articular Branch Block)
  Arms: Articular Branch Block (ABB)

SUMMARY:
Arthroscopic hip surgeries are increasingly being performed as both diagnostic and therapeutic interventions. These procedures are considerably painful, thus requiring the proper pain management techniques in order to provide patient satisfaction and sufficient pain control. Articular branch blocks have not been evaluated for their use in hip arthroscopy, but have potential advantages of blocking the sensory innervation of the entire hip joint, with minimal impact on motor innervation compared to alternative blocks.

This current study aims to evaluate the efficacy of using preoperative fluoroscopic-guided blockade of articular branches of the femoral and obturator nerves for analgesic management of patients undergoing arthroscopy compared to a saline sham block.

The utility of pre-operative hip articular branch block (ABB) prior to hip arthroscopy will provide superior pain management postoperatively compared to a saline sham block. We hypothesize that the ABB (Articular Branch Block) will reduce the area under the NRS pain scores by time curve (AUC) and decreased oral opioid milligram equivalent use in the first 24 hours post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for Hip Arthroscopy (Diagnostic or Therapeutic)
* Pre-operative Numeric Rating Score (NRS) for pain <8 on a 0 to 10 scale where 0 is no pain and 10 is worst pain imaginable.

Exclusion Criteria:

* Allergies to any of the study medications
* Anti-coagulation status (INR > 1.1, PT or APTT > 1.5 control)
* History of Hip Arthroplasty
* Infection of Hip
* Evidence of tumor
* Pregnancy
* History of diabetes with HbA1c > 10%
* Prior history of Hip Articular Branch Blockade or Hip Articular Branch PRF Ablation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
NRS Pain Scores (NRS) | 24 hours post-operatively
  Numerical Rating Scale is a self-reported pain assessment, in which a patient indicates their current pain level experienced. Patients can rate their pain on a scale of 0 (no pain) to 10 (worse pain imaginable). Higher scores indicated on this scale may indicate that a patient is experiencing higher pain intensities at that particular point in time. Whereas lower reported scores indicate that the patient is experiencing less intense or minimal pain.

SECONDARY OUTCOMES:
The QOR-15 (Quality of Recovery) | 24 hours post-operatively
  Quality of Recovery scores will be obtained 24 hours post-operatively. Scores are reported on an 11 point scale (0 to 10), where 0 = none of the time and 10 = all of the time. Higher scores indicated on the Quality of Recovery scale represent a better recovery outcome.
Analgesic medication use | 24 hours post-operatively

REFERENCES:
- [Background] Colvin AC, Harrast J, Harner C. Trends in hip arthroscopy. J Bone Joint Surg Am. 2012 Feb 15;94(4):e23. doi: 10.2106/JBJS.J.01886. PMID 22336982
- [Background] Yu HC, Al-Shehri M, Johnston KD, Endersby R, Baghirzada L. Anesthesia for hip arthroscopy: a narrative review. Can J Anaesth. 2016 Nov;63(11):1277-90. doi: 10.1007/s12630-016-0718-7. Epub 2016 Aug 16. PMID 27530361
- [Background] Steinhaus ME, Rosneck J, Ahmad CS, Lynch TS. Outcomes After Peripheral Nerve Block in Hip Arthroscopy. Am J Orthop (Belle Mead NJ). 2018 Jun;47(6). doi: 10.12788/ajo.2018.0049. PMID 29979805
- [Background] GARDNER E. The innervation of the hip joint. Anat Rec. 1948 Jul;101(3):353-71. doi: 10.1002/ar.1091010309. No abstract available. PMID 18873153
- [Background] Aprato A, Giachino M, Masse A. Arthroscopic approach and anatomy of the hip. Muscles Ligaments Tendons J. 2016 Dec 21;6(3):309-316. doi: 10.11138/mltj/2016.6.3.309. eCollection 2016 Jul-Sep. PMID 28066735
- [Background] Byrd JW. Hip arthroscopy. J Am Acad Orthop Surg. 2006 Jul;14(7):433-44. doi: 10.5435/00124635-200607000-00006. No abstract available. PMID 16822891
- [Background] Philippi MT, Kahn TL, Adeyemi TF, Maak TG, Aoki SK. Extracapsular local infiltration analgesia in hip arthroscopy patients: a randomized, prospective study. J Hip Preserv Surg. 2018 Sep 18;5(3):226-232. doi: 10.1093/jhps/hny030. eCollection 2018 Aug. PMID 30393549
- [Background] Kay J, de Sa D, Memon M, Simunovic N, Paul J, Ayeni OR. Examining the Role of Perioperative Nerve Blocks in Hip Arthroscopy: A Systematic Review. Arthroscopy. 2016 Apr;32(4):704-15.e1. doi: 10.1016/j.arthro.2015.12.022. Epub 2016 Feb 20. PMID 26907370
- [Background] Kapural L, Jolly S, Mantoan J, Badhey H, Ptacek T. Cooled Radiofrequency Neurotomy of the Articular Sensory Branches of the Obturator and Femoral Nerves - Combined Approach Using Fluoroscopy and Ultrasound Guidance: Technical Report, and Observational Study on Safety and Efficacy. Pain Physician. 2018 May;21(3):279-284. PMID 29871372
- [Background] Nye ZB, Horn JL, Crittenden W, Abrahams MS, Aziz MF. Ambulatory continuous posterior lumbar plexus blocks following hip arthroscopy: a review of 213 cases. J Clin Anesth. 2013 Jun;25(4):268-74. doi: 10.1016/j.jclinane.2012.11.013. Epub 2013 May 9. PMID 23665305
- [Background] Dold AP, Murnaghan L, Xing J, Abdallah FW, Brull R, Whelan DB. Preoperative femoral nerve block in hip arthroscopic surgery: a retrospective review of 108 consecutive cases. Am J Sports Med. 2014 Jan;42(1):144-9. doi: 10.1177/0363546513510392. Epub 2013 Nov 27. PMID 24284048
- [Background] Krych AJ, Baran S, Kuzma SA, Smith HM, Johnson RL, Levy BA. Utility of multimodal analgesia with fascia iliaca blockade for acute pain management following hip arthroscopy. Knee Surg Sports Traumatol Arthrosc. 2014 Apr;22(4):843-7. doi: 10.1007/s00167-013-2665-y. Epub 2013 Sep 24. PMID 24061718
- [Background] Lee EM, Murphy KP, Ben-David B. Postoperative analgesia for hip arthroscopy: combined L1 and L2 paravertebral blocks. J Clin Anesth. 2008 Sep;20(6):462-5. doi: 10.1016/j.jclinane.2008.04.012. PMID 18929290
- [Background] Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain. 2004 Sep-Oct;20(5):309-18. doi: 10.1097/00002508-200409000-00005. PMID 15322437
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Griffin DR, Parsons N, Mohtadi NG, Safran MR; Multicenter Arthroscopy of the Hip Outcomes Research Network. A short version of the International Hip Outcome Tool (iHOT-12) for use in routine clinical practice. Arthroscopy. 2012 May;28(5):611-6; quiz 616-8. doi: 10.1016/j.arthro.2012.02.027. PMID 22542434
- [Background] YaDeau JT, Tedore T, Goytizolo EA, Kim DH, Green DS, Westrick A, Fan R, Rade MC, Ranawat AS, Coleman SH, Kelly BT. Lumbar plexus blockade reduces pain after hip arthroscopy: a prospective randomized controlled trial. Anesth Analg. 2012 Oct;115(4):968-72. doi: 10.1213/ANE.0b013e318265bacd. Epub 2012 Jul 19. PMID 22822195